CLINICAL TRIAL: NCT00562705
Title: Effects of Growth Hormone Treatment on Eating Regulation and Comparison Between the Growth Responses With or Without Nutritional Intervention in Short Stature Children
Brief Title: Effects of Growth Hormone (GH) Treatment on Eating Regulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: rmc004623ctil
Record Dates: First submitted 2007-11-21; First posted 2007-11-22 (Estimated); Last update posted 2013-07-16 (Estimated); Status verified 2013-07

CONDITIONS: Short Stature
Keywords: growth hormone; eating regulation; nutritional intervention; short stature; ISS; SGA; IGHD; MPHD
MeSH Terms: conditions — Dwarfism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Growth hormone and nutritional intervention
  Interventions: Behavioral: growth hormone- Genotropin or NorditropinSimplex and nutritional intervention
- 2 (Active Comparator): growth hormone
  Interventions: Behavioral: growth hormone-Genotropin or NorditropinSimplex or "Biotropin"

INTERVENTIONS:
Behavioral: growth hormone- Genotropin or NorditropinSimplex and nutritional intervention — A combined treatment of growth hormone (Genotropin or NorditropinSimplex or "Biotropin") and nutritional intervention
  Arms: 1
Behavioral: growth hormone-Genotropin or NorditropinSimplex or "Biotropin" — Growth hormone treatment (Genotropin, or NorditropinSimplex or "Biotropin").
  Arms: 2

SUMMARY:
This is a two arm, randomized, prospective, intervention study in order to determine the effects of growth hormone treatment on eating regulation and to compare between the growth responses with or without nutritional intervention in short stature children.

The study will include 30 short stature children that are about to initiate growth hormone treatment and will last for one year. After 4 months of treatment, children will be randomized into two groups:

1. Control group that will continue with growth hormone treatment without any other intervention.
2. Study group that will be a given a nutritional intervention in addition to growth hormone treatment.

At screening visit and during the study the following parameters will be evaluated: height, weight, growth markers in the blood and urine, child eating behavior questionnaire, blood tests, hormonal tests and resting energy expenditure measurements.

DETAILED DESCRIPTION:
This is a two arm, randomized, prospective, intervention study in order to determine the effects of growth hormone treatment on eating regulation and to compare between the growth responses with or without nutritional intervention in short stature children.

Background:

In the last three decades children with different kinds of short stature pathologies were treated with growth hormone. Most of the attention in growth hormone studies is focused on the effect of the treatment on growth. Today there are very few studies that are focused on the effect of growth hormone on eating regulations and the connection between eating regulations and growth improvement in growth hormone treatment.

Objectives:

1. To evaluate the effect of short term growth hormone treatment on the following parameters:

   1. Appetite, food preference, amount of food and ingredients.
   2. Changes in food regulations.
   3. Changes in body composition.
   4. Changes in resting energy expenditure.
   5. Changes in hormones that are associated with appetite and with energy balance: IGF-1,IGFBP1&3 and Ghrelin.
   6. Changes in metabolic and nutritional measurements: glucose, insulin, lipid profile, total proteins, albumin, liver functions, alkaline-phosphatase, hemoglobin, transferrin, iron, B12, folic acid.
2. To evaluate the effect of nutritional support on growth rate in one year growth hormone treatment.
3. To evaluate changes in growth markers in the serum and urine during growth hormone treatment.

Methods:

The study will include 30 short stature children that are about to initiate growth hormone treatment and will last for one year. After 4 months of treatment children will be randomized into two groups:

1. Control group that will continue with growth hormone treatment without any other intervention.
2. Study group that will be given a nutritional intervention In addition to growth hormone treatment.

The nutritional intervention will include nutritional consultation and applying a personal dietetic menu. At screening visit and during the study the following parameters will be evaluated: height, weight, growth markers in the blood and urine, food diary, child eating behavior questionnaire, resting energy expenditure measurements, blood tests, hormonal tests and fasting and post-prandial levels of leptin, ghrelin, GLP-1, insulin and glucose.

ELIGIBILITY:
Inclusion Criteria:

1. Height of at least 2.0 standard deviations below the mean height for chronological age and sex according to the 2000 standards from the Centers for Disease Control and Prevention (CDC).
2. Children that have one of the following short stature pathologies:

   1. IGHD or MPHD
   2. ISS
   3. SGA
3. Proper function of thyroid gland, kidney and liver
4. Prior to initiating growth hormone treatment

Exclusion Criteria:

1. Chronic diseases
2. Diseases in the digestive system.
3. Neurological diseases.
4. Malignant diseases in the past or in the present. Treated with chemotherapy or radiation.
5. Genetic syndromes
6. Bone diseases
7. Taking chronic medicine, SSRI type, that effect the appetite and the growth hormone signal transduction.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 32 (Actual)
Dates: Start 2008-01; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
height and weight | every visit until the end of study
Growth markers | At screening visit, baseline and at the end of the visit

SECONDARY OUTCOMES:
Safety laboratory parameters | at screening, baseline and at the end of the study
food diary | every visit until the end of the study
Resting energy expenditure measurements | Every visit other than visit number 4

CONTACTS AND LOCATIONS:
Overall Officials: Moshe Phillip, Professor, Principal Investigator — Schneider Children Medical Center
Locations (1):
- Schneider Children's Medical Center, Petah Tikva, Israel